CLINICAL TRIAL: NCT04695444
Title: Comparison of the Effect of Tube Type and Intubation Technique on Nasopharyngeal Passage During Nasotracheal Intubation
Brief Title: Effect of Different Nasotracheal Tubes on Tube Passage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Chul Ho Chang, Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3-2020-0444
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Sialolithiasis
Keywords: nasotracheal intubation
MeSH Terms: conditions — Salivary Gland Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional PVC tube (Active Comparator): When performing nasotracheal intubation, clinicians use the conventional PVC tube.
  Interventions: Device: nasotracheal tube (Ring-Adair-Elwin)
- PVC tube with rubber suction catheter (Experimental): When performing nasotracheal intubation, clinicians use the conventional PVC tube + rubber suction catheter.
  Interventions: Device: nasotracheal tube (Ring-Adair-Elwin)
- velvet soft PVC tube (Experimental): When performing nasotracheal intubation, clinicians use the velvet soft PVC tube.
  Interventions: Device: nasotracheal tube (portex)

INTERVENTIONS:
Device: nasotracheal tube (Ring-Adair-Elwin) — different materials for nasotracheal intubation conventional PVC tube
  Other Names: nasal RAE (Ring-Adair-Elwin) tube
  Arms: conventional PVC tube
Device: nasotracheal tube (Ring-Adair-Elwin) — different materials for nasotracheal intubation conventional PVC tube with rubber suction catheter
  Other Names: nasal RAE (Ring-Adair-Elwin) tube
  Arms: PVC tube with rubber suction catheter
Device: nasotracheal tube (portex) — different materials for nasotracheal intubation velvet soft PVC tube.
  Other Names: portex tube
  Arms: velvet soft PVC tube

SUMMARY:
The purpose of the study is to find out the clinical effects that can be obtained during nasotracheal intubation when using velvet-soft PVC tube compared to conventional polyvinylchloride(=PVC) tube.

DETAILED DESCRIPTION:
The hypothesis of this study is that the velvet-soft PVC tube can advanced from the nasal cavity to the oral cavity through the posterior wall of the pharynx more smoothly than conventional PVC tube, thus reducing blockade of tube advancement, nasal/pharyngeal mucosal bleeding, and intubation time. In addition, investigators would like to compare the technique of nasal intubation using by connecting rubber suction catheter to PVC tube tip.

ELIGIBILITY:
Inclusion Criteria:

* The patients who need to nasotracheal intubation for surgery
* age: 19 years old or more

Exclusion Criteria:

* patient refusal
* nasal deformity
* history of previous moderate degree of epistaxis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
blockade of tube advancement from the nasal cavity to the oral cavity [ during intubation] | During nasotracheal intubation (From the time of insertion of the tube through the nostril to completion of the intubation )
  When entering a nasotracheal tube from the nasal cavity to the oral cavity before use of laryngoscope in nasotracheal intubation, clinicians sometimes encounter blockade of in tube advancement. The reason is that the direction of the nasotracheal tube and the posterior wall of the nasopharynx are anatomically perpendicular. When advancing the tube from the nasal cavity to the oral cavity, the researcher will evaluate the presence of blockade of tube advancement in the pharynx. (none / present)

SECONDARY OUTCOMES:
Intubation time | During nasotracheal intubation (From the time of insertion of the tube or tube combined with the rubber suction catheter to the completion of nasotracheal intubation)
  the total time of nasotracheal intubation: From the time of insertion of the tube or tube combined with the rubber suction to the completion of nasotracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Chul Ho Chnag, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Kim H, Lee JM, Lee J, Hwang JY, Chang JE, No HJ, Won D, Row HS, Min SW. Effect of neck extension on the advancement of tracheal tubes from the nasal cavity to the oropharynx in nasotracheal intubation: a randomized controlled trial. BMC Anesthesiol. 2019 Aug 17;19(1):158. doi: 10.1186/s12871-019-0831-6. PMID 31421677
- [Derived] Lee J, Lee JM, Shim YH, Cho JG, Lee J, Lim JY, Chang CH. A randomized comparison of three intubation techniques/tube materials for nasotracheal intubation. Can J Anaesth. 2024 Jul;71(7):978-986. doi: 10.1007/s12630-024-02743-z. Epub 2024 Mar 28. PMID 38548948